CLINICAL TRIAL: NCT03546569
Title: Circulation Tumor Cells, Tumor DNA and Immunological Response in Relation to Colonic Stent Placement for Malignant Obstruction
Brief Title: Tumor Cells, Tumor DNA and Immunological Response in Colonic Stent Placement
Acronym: CISMO
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-059-2017
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Cancer of Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate levels of circulating cell free DNA (cfDNA), circulating tumor DNA (ctDNA), circulating tumor cells (CTC) and immunological changes after self-expanding metal stent (SEMS) placement for malignant obstruction in the colon, and interpret these levels in relation to overall- and disease-free survival.

Furthermore, we intend to study the opportunity to identify patients with a higher risk of recurrence due to the SEMS placement by monitoring cfDNA and ctDNA-levels, as it may be a potential biomarker to initiate or optimize chemotherapy and thereby ensure a better prognosis for the patients.

DETAILED DESCRIPTION:
Study design This prospective study will include 20 patients undergoing SEMS placement as a bridge to elective surgery at Koege- and Slagelse Hospital. Baseline blood samples will be collected before the procedure. After the procedure blood samples will be collected 1, 4, 12 and 24 hours after SEMS placement. After elective surgery a tumor sample will be collected.

Prior to SEMS placement:

When potential candidates are admitted to the hospital they will be presented to the study by the relevant surgeon. The investigators will be contacted, when the patient is admitted to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 to 95 years
* Patients with acute malignant obstruction in the colon.
* ASA class I-III (Classification of the American Society of Anesthesiology)
* Signed informed consent

Exclusion Criteria:

* Known immune-defects
* Withdrawal of informed consent
* Bloodtransfusion 24 hours prior to stent-placement until 24 hours after stent-placement.
* Surgery within 24 hours after stent-placement
* Known inflammatory bowel disease

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We intend to include 20 patients with malignant obstruction who are treated with a colorectal stent as bridge to surgery or as palliation.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
ctDNA/cfDNA levels in relation to colorectal stent placement | 2 years
  Blood samples will be collected before the treatment and again 1, 4, 12 and 24 hours after stent placement.

SECONDARY OUTCOMES:
Immunological response | 2 years
  Flow cytometry will be performed and additionally multiplex cytokine analyses will be performed
Metastatic ability of the cancer cells | 2 years
  Cell adhesion assay, proliferation and migration will be performed on serum.

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Køge, Denmark